CLINICAL TRIAL: NCT06587802
Title: Phase II Study of PD-1 Antibody Combined With Radiotherapy in Recurrent or Metastatic Adrenal Cortical Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Director, Head of urology, Principal Investigator, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2024-545-01
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenocortical Carcinoma; radiotherapy; immunotherapy
MeSH Terms: conditions — Adrenocortical Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): SBRT radiotherapy (radiotherapy dose: 40Gy, 5 times, 8Gy each time, number of metastatic radiotherapy: ≤5).At the end of radiotherapy, 240mg of triplizumab was administered intravenously every cycle (21 days)
  Interventions: Drug: Triprolizumab; Device: rodiotherapy

INTERVENTIONS:
Drug: Triprolizumab — At the end of radiotherapy, 240mg of triplizumab was administered intravenously every cycle (21 days)
Device: rodiotherapy — SBRT radiotherapy (radiotherapy dose: 40Gy, 5 times, 8Gy each time, number of metastatic radiotherapy: ≤5)

SUMMARY:
Adrenal cortical cancer is an extremely rare and highly aggressive malignancy with an incidence of 0.7-2 per million people · year and a 5-year overall survival rate of 15-44%, among which the 5-year survival rate of stage IV cortical cancer is only 13% and the prognosis is poor. Complete surgical resection is one of the most important ways to cure cortical cancer, but the surgical trauma is large, the complications are high, the postoperative recovery of patients is slow, and the tumor is difficult to achieve complete resection, and the postoperative recurrence and metastasis rate of patients is high, even for localized cortical cancer (stage I-III), the recurrence and metastasis rate is still close to 60%.

Recurrent or metastatic cortical cancer is mainly treated with drugs. However, the current first-line drug therapy is only 22.3% effective, the tumor progression-free time is 5.6 months, and the serious adverse reaction rate is as high as 58.1%.

The effective rate of second-line treatment with chemotherapy and targeted drugs was less than 10%, and the tumor progression-free time was only 2.8 months.

The Phase II study of PD-1 monoclonal antibody in the treatment of cortical cancer showed that the treatment effective rate was 23%, and the tumor progression-free survival time was 2.1 months, which was comparable to the first-line regimen, and has been approved by the guidelines for advanced cortical cancer.

Radiation therapy has high efficiency and local control rate, small side effects, and can inhibit tumor growth, relieve local pressure and pain. However, it only has a good effect on the irradiated site, and it is difficult to inhibit the progression of non-radiotherapy lesions and the generation of other new lesions.

The synergistic effect of immunotherapy combined with radiation therapy for metastatic stoves has been confirmed in many solid tumors such as kidney cancer, which can improve the local control rate of solid tumors and prolong the time of tumor progressive-free.

In the early stage, this research team applied PD-1 monoclonal antibody combined with radiotherapy to treat recurrent or metastatic adrenal cortical cancer in many cases after receiving first-line drug therapy regimen, which not only achieved local control of the radiotherapy focus, but also inhibited the progression of other metastases, and achieved longer disease control effect.

DETAILED DESCRIPTION:
Adrenocortical Carcinoma (ACC) is an extremely rare and highly aggressive malignant tumor with an incidence of 0.7-2 per million people and poor prognosis. The 5-year overall survival rate is 15-44%, and the 5-year survival rate of stage IV ACC is only 13%. Surgical complete resection (R0) is one of the most important ways to cure ACC. However, even for localized ACC (stage I-III), there is still a recurrence and metastasis rate of nearly 60%, due to reasons including surgical failure to achieve R0 resection, tumor rupture, and postoperative hematologic and lymphatic metastasis. Recurrent or metastatic ACC is mainly treated with systemic drugs, mitotan monotherapy or mitotan combined with cisplatin based chemotherapy (mitotan ± etoposide, adriamycin and cisplatin: EDP-M protocol is currently the first-line protocol for advanced ACC, but the objective response rate (ORR) of EDP-M is only 22.3%, the progression-free survival (PFS) is 5.6 months, and the grade 3-4 adverse reactions are as high as 58.1%. Treatment options for patients with recurrent or metastatic ACC after first-line treatment progress are more limited and less effective. The ORR of second-line chemotherapy for advanced ACC was less than 10%. Targeted drugs such as Sunitinib for second-line treatment of advanced ACC had an ORR of 0, and PFS was only 2.8 months. Five clinical studies have been conducted to investigate the efficacy of immunotherapy for adrenal cortical cancer. The results of a phase II study on the treatment of ACC with PD-1 monoclonal antibody showed that ORR could reach 23%, which is the regimen with the highest objective response rate at present. Therefore, the guidelines recommend PD-1 monoclonal antibody for advanced ACC, but the PFS of PD-1 monoclonal antibody is only 2.1 months. Therefore, how to prolong PFS with high ORR is a difficult problem in the treatment of advanced ACC.

For recurrent or metastatic ACC, surgical palliative resection of metastasis can reduce tumor or alleviate symptoms. However, due to large surgical trauma, high complications, slow postoperative recovery of patients, difficult R0 resection of tumors, and high postoperative recurrence and metastasis rate of patients, it is still controversial whether palliative surgery for advanced ACC can bring survival benefits to patients. The guidelines also recommend that radiotherapy can be used for advanced ACC, with high ORR and local control rate, small side effects, inhibiting tumor growth, relieving local pressure and pain. However, radiotherapy is a local treatment that only has a good effect on the irradiated site, and it is difficult to inhibit the progression of non-radiotherapy lesions and the emergence of other new lesions. Therefore, the effect of radiotherapy alone on the overall disease control of patients with advanced ACC recurrence or metastasis is still unsatisfactory.

The synergistic effect of immunotherapy combined with radiotherapy for metastatic stoves has been demonstrated in many solid tumors such as kidney cancer. The ORR of advanced renal clear cell carcinoma treated with PD-1 monoclonal antibody alone was only 36.5%, the median PFS time was 7.1 months, and the 2-year PFS rate was 22.3%, while the ORR of advanced renal clear cell carcinoma treated with PD-1 monoclonal antibody combined with radiotherapy was 63%, PFS was 15.6 months, and the 2-year PFS rate was 45%. Therefore, immunotherapy combined with radiotherapy can improve the local control rate and prolong the PFS time of metastatic renal carcinoma. The ORR of PD-1 monoclonal antibody monotherapy for advanced ACC was 23% and PFS was 2.1 months. Although the ORR was similar to that of EDP-M first-line regimen, the PFS was shorter. Therefore, it is of great clinical significance to explore whether PD-1 monoclonal antibody combined with radiotherapy for advanced ACC can obtain higher ORR and longer PFS.

In the early stage, this research team applied PD-1 monoclonal antibody combined with SBRT to treat recurrent or metastatic adrenal cortical cancer in multiple cases of recurrent or metastatic ACC after treatment with first-line EDP-M protocol, which not only achieved local control of radiotherapy lesions, but also inhibited the progression of other metastasies, and achieved longer disease control effect (ORR: 4/7, PFS: July). On the basis of previous practice, our team plans to further conduct prospective exploratory clinical research on the efficacy and safety of PD-1 monoclonal antibody combined with radiotherapy in the treatment of recurrent or metastatic adrenal cortical carcinoma, so as to provide more safe and effective treatment options for this rare tumor.

Main purpose:

To observe and evaluate the progression-free survival time of PD-1 monoclonal antibody combined with radiotherapy in the treatment of recurrent or metastatic adrenal cortical carcinoma

Secondary purpose:

To observe and evaluate the secondary efficacy indexes and safety of PD-1 monoclonal antibody combined with radiotherapy in the treatment of recurrent or metastatic adrenal cortical carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participated in this study and signed informed consent;
* Patients ≥18 years old;
* ECOG score ≤2 points; Expected survival ≥6 months;
* Pathological diagnosis of adrenal cortical carcinoma;
* Inability or unwillingness to surgically resect recurrent or metastatic adrenal cortical cancer;
* Adrenal cortical cancer has recurred or metastasized after receiving mitotan monotherapy, chemotherapy, or first-line regimens based on mitotan combined with cisplatin chemotherapy and has progressed, unable to tolerate or unwilling to accept the regimens;
* Have at least one measurable lesion (RECIST1.1);
* The main organs function well, and the laboratory examination indicators meet:
* (1) Blood routine examination: Hemoglobin (HB) ≥90g/L(5.6mmol/L); Absolute neutrophil count (ANC) ≥1.5×109/L; Total white blood cells ≥3.5×109/L;

  * Platelet (PLT) ≥80×109/L; (2) Blood biochemical examination:

    ① Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (liver metastasis/bone metastasis ≤5× ULN; Tumor bone metastasis ≤5ULN);

    ② Serum total bilirubin (TBIL) ≤1.5×ULN;
  * Serum creatinine Cr≤1.5×ULN or creatinine clearance ≥60ml/min; Blood urea nitrogen (BUN)≤2.5× upper limit of normal value (ULN); ④ Albumin (ALB)≥30g/L; (3) Blood coagulation test: Activated partial thromboplastin time (APTT), International Normalized ratio (INR), prothrombin time (PT) ≤1.5×ULN;
* Women of childbearing age must confirm their non-pregnant status before enrollment, and all enrolled subjects (whether male or female) should take adequate contraceptive measures during the whole treatment period and 4 weeks after the end of treatment;
* The subjects were willing to return to the hospital for follow-up and had good compliance.

Exclusion Criteria:

* Receiving anti-tumor monoclonal antibodies or other investigational drugs before enrollment
* Previously received other anti-PD-1 monoclonal antibody therapy or other drug therapy for PD-1 / PD-L1
* Radiotherapy has been used in the lesion area in the past
* The lesion invades the intestinal duct, and there are contraindications to radiotherapy such as the risk of intestinal fistula caused by radiotherapy
* Known allergic reaction to the active ingredient of PD-1 monoclonal antibody or any excipients
* Have a medical condition that interferes with oral medication, including but not limited to difficulty swallowing, chronic diarrhea, or intestinal obstruction
* Uncontrolled heart disease, such as heart failure with NYHA rating ≥2, unstable angina pectoris, history of myocardial infarction in the past year, and ventricular or supraventricular arrhythmias requiring treatment
* Central nervous system metastasis with clinical symptoms, such as brain edema, requiring hormonal intervention, or brain metastasis progression;
* Serious infections (CTCAE > Grade 2) occurred within 4 weeks prior to the first use of the study drug, such as severe pneumonia, bacteremia, and infection complications requiring hospitalization; Baseline chest imaging examination indicating active lung inflammation, signs and symptoms of infection within 2 weeks prior to first use of the study drug, or the need for oral or intravenous antibiotic treatment (excluding prophylactic antibiotic use)
* Receive systemic sex hormone or other immunosuppressive therapy with an equivalent dose greater than 10mg prednisone/day within 4 weeks of signing the informed consent. Participants with a systemic sex hormone dose ≤10mg prednisone/day or inhaled/topical corticosteroids could be enrolled
* chronic hepatitis B active stage or active hepatitis C patients. Screening period hepatitis B surface antigen (HepatitsBSurfaceAntigen, HBsAg) or hepatitis b core antibody (HBcAb HepatitsBcoreAntibody,) or hepatitis c virus (HepatitisCVirus, HCV) antibody positive patients, Only through HepatitisBVirus (HBV) DNA detection (no more than 104 copies /mL or 2000IU/mL) and HCVRNA detection (no more than the lower limit of the assay) will he be included in the group test after the disease has been controlled. Hepatitis B virus carriers, hepatitis B whose disease has been controlled after drug treatment (no more than 104 copies /mL of DNA or 2000IU/mL), and cured hepatitis C patients can be enrolled
* Significant vital organ dysfunction or uncontrollable comorbiditions, including but not limited to uncontrolled hypertension, decompensated cirrhosis, active peptic ulcer or bleeding disease
* History of interstitial lung disease or non-infectious pneumonia; Participants with a history of drug-induced or radiation-induced non-infectious pneumonia without symptoms were admitted
* Pregnant and lactating women and subjects of childbearing age who do not want to take contraceptive measures
* Persons with mental illness, a history of alcohol or drug abuse, or inability to obtain informed consent
* Other researchers have determined that participants are not suitable for this study, such as serious diseases, including mental illness, serious abnormal test results, and other social or family high-risk risk factors that require timely intervention
* refuse or can not sign the informed consent.
* Patients suspected of having other primary cancers; Patients with other primary malignancies within the 5 years prior to the study period (other than adequately treated cervical or skin cancer in situ, such as basal cell carcinoma, squamous cell carcinoma, or non-melanoma skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2027-03-14 (Estimated); Study Completion 2027-03-14 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From study enrollment to the time of tumor progression, at least 3 year follow-up

SECONDARY OUTCOMES:
Overall survival time | From study enrollment to the end of treatment or death up to 4 years follow-up
Duration of remission | From complete or partial response of tumor to the end of tumor progression or death, at least 3 year follow-up
Objective response rate | From study enrollment to the end of complete response or partial response of tumor, at least 3 year follow-up
Duration of remission | From partial response or completed response of tumor to the end of tumor progression or death, at least 3 years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Research Data Deposit ：https://www.researchdata.org.cn/
Supporting Information: Study Protocol, SAP
URL: https://www.researchdata.org.cn/